CLINICAL TRIAL: NCT02972281
Title: Systematic Search for Primary Immunodeficiency in Adults With Unexplained Recurrent and/or Severe Infections With Encapsulated Bacteria
Brief Title: Systematic Search for Primary Immunodeficiency in Adults With Infections
Acronym: SPIDAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: deficient inclusions
Sponsor: University Hospital, Lille (Other)
Collaborators: Imagine Institute (Other); Octapharma (Industry); CSL Behring (Industry); Laboratoire français de Fractionnement et de Biotechnologies (Industry); Air Liquide SA (Industry); The Binding Site Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014_07; 2014-A00739-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Complement Deficiency; Antibody Deficiency; Chronic Sinus Infection; Meningitis, Bacterial; Pneumonia, Bacterial; Otitis Media; Streptococcal Infection; Neisseria Infections; Haemophilus Influenza; Pneumococcal Infections
MeSH Terms: conditions — Hereditary Complement Deficiency Diseases; Meningitis, Bacterial; Pneumonia, Bacterial; Otitis Media; Streptococcal Infections; Pneumococcal Infections | interventions — Immunologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with bacterial infections (Other): Patients with recurrent and/or severe bacterial infections
  Interventions: Biological: Immunological diagnosis tests

INTERVENTIONS:
Biological: Immunological diagnosis tests — (Non exhaustive list): hemogram, IgG, A, M, IgG subclasses, complement, vaccinal response to protein and polysaccharide antigens, ...

SUMMARY:
Antibody deficiencies and complement deficiencies are the most frequent Primary immunodeficiencies (PIDs) in adults, and are associated with greatly increased susceptibility to recurrent and/or severe bacterial infections - especially upper and lower respiratory tract infections and meningitis. The literature data suggest that PIDs are under-diagnosed in adults. The current European and US guidelines advocate screening adults for PIDs if they present recurrent benign especially upper and lower respiratory tract infections, or if they have experienced at least two severe bacterial infections and/or have a recurrent need for intravenous antibiotics. The objective of the demonstrate the interest of PIDs screening in adult patients who present such recurrent infections and/or after the first severe bacterial infection, especially when the patients do not present with known, etiologically relevant comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yrs old patients
* ≥ 2 bacterial upper or lower respiratory tract infections/years, for at least 2 years, or
* ≥ 1 severe bacterial upper or lower respiratory tract infection requiring hospitalization and IV antibiotics, or
* ≥ 1 invasive infection (meningitis, bacteriemia, arthritis) due to Streptococcus pneumoniae, group A Streptococcus, Haemophilus influenzae, Neisseria meningitidis or Neisseria gonorrhoeae

Exclusion Criteria:

* concomitant, systemic comorbidity that predisposes to infection (solid or hematological cancer, diabetes mellitus, severe alcohol or intravenous drug abuse, chronic liver or kidney failure, human immunodeficiency virus infection, anatomic or functional asplenia, drug-induced 1 neutropenia, or solid organ or hematopoietic stem cell transplantation).
* the presence of a local predisposing factor: cigarette smoking (> 5 pack-year and/or 5 cigarettes/day), underlying infection (tuberculosis, influenza…), chronic obstructive pulmonary disease, cystic fibrosis or bronchiectasis for pulmonary infections; cerebrospinal leak or preceding upper respiratory tract (URT) infections for non-meningococcal meningitis; oral, dental or skin condition for GAS infections
* use of corticosteroids, non-steroidal anti-inflammatory drugs, immunosuppressants or cytotoxic chemotherapeutics
* PID diagnosed before the infectious episode in question.
* current or recent pregnancy
* hospital-acquired infection (including infections of prostheses).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Frequency of Primary immunodeficiencies (PIDs) in adult patients with recurrent and/or severe bacterial infection with encapsulated bacteria | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lefevre, MD, Principal Investigator — University Hospital, Lille
Locations (19):
- France (19):
  - Ch Armentieres, Armentières
  - CH ARRAS, Arras
  - Ch Bethune, Béthune
  - Ch Boulogne-Sur-Mer, Boulogne-sur-Mer
  - Ch Cambrai, Cambrai
  - Ch Denain, Denain
  - CH DOUAI, Douai
  - Ch Dunkerque, Dunkirk
  - CH LENS, Lens
  - Hopital Prive La Louviere, Lille
  - CHRU,, Lille
  - Hopital Saint Vincent - Saint Antoine, Lille
  - Ch Arrondissement de Montreuil, Rang-du-Fliers
  - C.H de Roubaix, Roubaix
  - Ch Region de St-Omer, Saint-Omer
  - Groupe Hospitalier Seclin Carvin, Seclin
  - Ch Tourcoing, Tourcoing
  - Ch de Valenciennes, Valenciennes
  - Clinique Teissier, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stabler S, Lamblin C, Gaillard S, Just N, Mihailescu M, Viget N, Sy Ndiaye T, Dzeing Ella A, Brunin G, Weyrich P, Prevotat A, Chenivesse C, Le Rouzic O, Mortuaire G, Vuotto F, Faure K, Leurs A, Wallet F, Loiez C, Titecat M, Le Guern R, Hachulla E, Sanges S, Etienne N, Terriou L, Launay D, Lopez B, Bahuaud M, Batteux F, Dubucquoi S, Gesquiere-Lasselin C, Labalette M, Lefevre G; DIPANOR network. High Frequency of Specific Polysaccharide Antibody Deficiency in Adults With Unexplained, Recurrent and/or Severe Infections With Encapsulated Bacteria. Clin Infect Dis. 2023 Mar 4;76(5):800-808. doi: 10.1093/cid/ciac842. PMID 36285530